CLINICAL TRIAL: NCT03650595
Title: MRI Guided Focal Laser Ablation of Prostate Cancer
Acronym: MRgFLA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Clinical Laserthermia Systems AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-9002
Record Dates: First submitted 2018-08-10; First posted 2018-08-28 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer; Low and Intermediate Risk Prostate Cancer
Keywords: MRI; Focal Laser Ablation; MR-Guided Focal Laser Ablation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: 24 Month, Prospective, Interventional, Open-label Single-Arm Effectiveness Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm prospective clinical trial (Experimental): This is a single arm study where patients with low-intermediate risk MR visible locally confined prostate cancer will be treated with focal laser ablation under MRI guidance in the magnet. Following treatment, the patients will be assessed by MRI and Biopsy at 6 months and at 2 years, with PSA assessment at regular intervals during the time
  Interventions: Device: The TRANBERGCLS|Thermal Therapy

INTERVENTIONS:
Device: The TRANBERGCLS|Thermal Therapy — MRI Guided Focal Laser Ablation of Prostate Cancer by The Diode Laser System - The TRANBERGCLS|Thermal Therapy

SUMMARY:
This clinical research study is designed to determine the ability of in bore MRI guided Focal Laser Ablation (MRgFLA) in patients with early stage carcinoma of prostate. The results will be evaluated by repeated MRI and prostate biopsy. Previous prospective development study demonstrated that FLA may be a viable option for men with low-intermediate risk prostate cancer. The vast majority of patients undergoing this treatment experienced minimal side effects with no peri-operative complications. Over 80% of patients treated with MRgFLA remain on AS and were able to avoid radical therapy at mean follow up duration of 3 years.

DETAILED DESCRIPTION:
Study Objectives are to evaluate the proportion of patients with low-intermediate risk prostate cancer undergoing focal laser ablation (MRgFLA) prostate treatment who will be free of clinically significant Prostate Cancer (PCa), when using a > 5mm margins around the MR visible tumor in defining the ablation contour. The rationale of the study is to show that MRgFLA is a safe procedure that can significantly postpone or eliminate the need for patients with Low-Intermediate Risk prostate cancer to undergo a definitive treatment (i.e., Radical Prostatectomy or Radiation therapy) for their disease. Study population: patients with Low-Intermediate Risk Prostate Cancer who are willing to take part in the study and meet study eligibility criteria. Primary Study Objective is to show that MRgFLA can significantly reduce the need for definitive treatment (e.g., Radical Prostatectomy, or Radiation therapy) and is a safe procedure for patients with Low-Intermediate Risk Prostate Cancer defined in the current protocol as 1) Gleason score 6 and 7 (=3+4 or 4+3; No Grade 5 pattern), and 2) T1-T2, N0, M0.

ELIGIBILITY:
Inclusion Criteria:

* Men 40-80 years of age
* Histologically proven low-intermediate risk prostate carcinoma; (Gleason score ≤ 7, primary grade ≤ 4;)
* Prostate cancer clinical stage T1c and T2
* MR site suspicious for cancer or cancer mapped to one lobe of the prostate using the 3D hybrid TRUS device
* Size of MR visible tumor <20mm
* Suspicious site on Prostate MRI must coincide with sector positive for cancer on biopsy
* Prostate specific antigen (PSA) level <15 ng/mL
* IPSS, ICIQ-UI-SF, IIEF complete prior to procedure
* Life expectancy of greater than 10 years, based on co-morbidity not related to prostate cancer.

Exclusion Criteria:

* Medically unfit for focal therapy of the prostate
* Patients who are unwilling or unable to give informed consent;
* Patients who have received androgen suppression therapy
* Patients who have received or are receiving chemotherapy for prostate carcinoma;
* Patients previously treated with surgery to the prostate (traditional, endoscopic or minimally invasive including HIFU, TUNA, RITA, microwave, cryotherapy or any curative treatment
* Patients who have undergone radiation therapy for prostate cancer or to the pelvis
* Any condition, or history of illness or surgery that, in the opinion of the Investigator, might confound the results of the study or pose additional risks to the patient (e.g. significant cardiovascular conditions or allergies);
* Patients with a history of noncompliance with medical therapy and/or medical recommendations;
* Patients who are unwilling or unable to complete the patient self-assessment questionnaires;
* Chronic or acute prostatitis, neurogenic bladder, urinary tract infection, sphincter abnormalities, or any other symptom that prevents normal micturition.
* Patients who have participated in a clinical study and/or received treatment with an investigational treatment and/or product within the past 90 days;
* Patients with contraindication to MRI (i.e. pacemaker, hip prosthesis, severe claustrophobia, brain aneurysm clip, allergy to MRI contrast agent)
* Any condition, or history of illness that, in the opinion of the investigator will confound or increase the patient risk during the study

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men with prostate cancer
Enrollment: 102 (Estimated)
Dates: Start 2018-03-29 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of study patients clinically free of clinically significant PCa (i.e. requires definitive treatment) | 6 months after treatment completion
  Clinically significant PCa will be defined as recurrent/residual Gleason 3+4 or higher, and/or high-volume Gleason 6 disease found at 6-month biopsy.
The proportion of study patients clinically free of clinically significant PCa (i.e. requires definitive treatment) | 24 months after treatment completion
  Clinically significant PCa will be defined as recurrent/residual Gleason 3+4 or higher, and/or high-volume Gleason 6 disease found at 24-month biopsy.

SECONDARY OUTCOMES:
Treatment effect on patients' Quality of Life (QoL), the following validated self-reported urogenital functioning assessment instruments will be used before and following treatment at pre-specified interval | Baseline before treatment, 30 days, 6 months, 12 months and at 24 months following treatment
  Validate Patient-Reported Questionnaire (International Prostate Symptom Score, scale from 0-7 mild, 8-19 moderate, 20-35 severe symptoms, higher values being worse, averages at different time points will be noted to assess improvement, decline or baseline) will be completed by participants throughout the study to assess Health Related Quality of Life.
Treatment effect on patients' Quality of Life (QoL), the following validated self-reported urogenital functioning assessment instruments will be used before and following treatment at pre-specified interval | Baseline before treatment, 30 days, 6 months, 12 months and at 24 months following treatment
  Validate Patient-Reported Questionnaire (International Index of Erectile Function-15, higher scores are better, averages at each specified interval will be taken once all subjects reach the interval and study completion) will be completed by participants throughout the study to assess Health Related Quality of Life.

CONTACTS AND LOCATIONS:
Overall Officials: Sangeet Ghai, MD, Principal Investigator — Director; Biopsy Centre, Abdominal Division and Joint Department of Medical Imaging
Locations (1):
- Sangeet Ghai, MD, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No